CLINICAL TRIAL: NCT02572648
Title: A Comparison of Magnetic Resonance Imaging in Persons With Heart Failure to Health, Aged Matched Controls (MIND-HF)
Brief Title: A Comparison of Magnetic Resonance Imaging in Persons With Heart Failure to Health, Aged Matched Controls
Acronym: MIND-HF
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Gary, Associate Professor, Emory University
Other Study IDs: IRB00083607
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
Keywords: Cardiomyopathy; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Participants with Heart Failure: Participants with heart failure will complete neurocognitive tests and undergo magnetic resonance imaging (MRI).
  Interventions: Other: Brain Imaging (Neuroimaging); Other: Cognitive Function Assessment
- Healthy Controls: Healthy controls will complete neurocognitive tests and undergo magnetic resonance imaging (MRI).
  Interventions: Other: Brain Imaging (Neuroimaging); Other: Cognitive Function Assessment

INTERVENTIONS:
Other: Brain Imaging (Neuroimaging) — Magnetic Resonance Imaging (MR) will be acquired on a research dedicated Siemens 3Tesla TIM TRIO MRI scanner with a 32-channel head coil.The MRI scanning protocol will have scans to measure voxelwise and whole-brain measures of grey matter (GM) volumes through a high resolution T1-weighted (T1W) multi-echo magnetization prepared gradient echo (MEMPRAGE) anatomic scan.
  Total time in scanner will be approximately 53 minutes.
Other: Cognitive Function Assessment — Cognitive function will be assessed using several batteries; the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), the Controlled Oral Word Association Test (COWA), the Color Trails 1 & 2, the WAIS-III Digit Span and Letter Number Sequence test, the Stroop Test, and the California Computerized Assessment Package Reaction Time test (CALCAP).

SUMMARY:
The purpose of this study is to examine the relation between the structural brain changes associated with heart failure, neurocognitive performance, and how these changes impact self-care behaviors.

DETAILED DESCRIPTION:
The purpose of this study is use neuroimaging techniques to better understand the underlying structural brain changes and physiological mechanisms that guide the thinking and decision making processes required for people with heart failure. The study will compare how the underlying brain structures and circulation are similar to or different in persons with heart failure to healthy, aged matched controls using special neuroimaging procedures.

ELIGIBILITY:
Inclusion Criteria:

Participants with heart failure:

* Speak and understand English
* Live independently within a 60 mile radius of Atlanta
* Montreal Cognitive Assessment (MOCA) score of less than or equal to 24
* Documented medical diagnosis of New York Heart Association (NYHA) class II or III systolic
* Left ventricular ejection fraction (LVEF) greater than or equal to 10% that is documented within the last year by echocardiogram, cardiac catheterization ventriculography, or radionuclide ventriculography
* Receiving medication therapy for heart failure (HF) according to American College of Cardiology (ACC) American Heart recommendation guidelines for at least 8 weeks prior to study enrollment

Healthy Controls

* Speak and understand English
* Live independently within a 60 mile radius of Atlanta

Exclusion Criteria:

Participants with heart failure:

* New York Heart Association (NYHA) class I or IV
* Change in heart failure (HF) therapy within 6 months
* Worsening of heart failure (HF) symptoms within last 5 days
* Unstable angina
* Renal insufficiency (serum creatinine greater than 3.o mg/dL)
* Hospitalized within the last 30-days
* Diagnosed with any neurological disorder that may interfere with cognitive function
* Beck Depression Inventory II (BDI-II) score greater than 25
* Claustrophobia
* Implanted devices such as internal cardiac defibrillator or pacemaker
* Carrying non-removable objects
* Stents
* Body weight more than 120 kg

Healthy Controls

* Taking prescription medications
* Cardiovascular disease;
* Cerebrovascular disease
* Neurological disease
* Respiratory disease
* Claustrophobia
* Any implanted metal objects not considered safe or appropriate for the MRI environment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women with heart failure and men and women without heart failure to serve as healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Structural White Matter | Visit 1 (Up to 2 hours)
  Diffusion tensor imaging (DTI) and myelin water imaging (MWI) will be used to compare brain structural white matter between participants with heart failure and healthy controls. This will be obtained via magnetic resonance imaging (MRI) techniques.

SECONDARY OUTCOMES:
Functional Connectivity | Visit 1 (Up to 2 hours)
  Functional connectivity that regulates neurocognitive functions will be assessed by blood oxygen level dependent resting state functional MRI (rsFMRI).This will be obtained via magnetic resonance imaging (MRI) techniques.
Global Cerebral Blood Flow (CBF) | Visit 1 (Up to 2 hours)
  Arterial spin labeling (ASL) based magnetic resonance (MR) perfusion imaging will evaluate global cerebral blood flow (CBF). This will be obtained via magnetic resonance imaging (MRI) techniques.
Regional Cerebral Blood Flow (CBF) | Visit 1 (Up to 2 hours)
  Arterial spin labeling (ASL) based magnetic resonance (MR) perfusion imaging will evaluate regional cerebral blood flow (CBF). This will be obtained via magnetic resonance imaging (MRI) techniques.
Structural Grey Matter | Visit 1 (Up to 2 hours)
  Voxel-based morphometry (VBM) of T1-weighted (T1w) high-resolution magnetic resonance imaging MRI anatomics will be used to measure brain structural white matter.
Cognitive Function assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Visit 2 (Up to 2 hours)
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a brief, individually administered test designed to evaluate neuropsychological status of adults, ages 20-89. The 12 subtests measure attention, language, visuospatial/constructional abilities, and immediate and delayed memory.
Cognitive Function assessed by the Controlled Oral Word Association (COWA) Test | Visit 2 (Up to 2 hours)
  The Controlled Oral Word Association (COWA) Test is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter. The more words produced in the allotted time period the higher the score.
Cognitive Function assessed by the Color Trails Test | Visit 2 (Up to 2 hours)
  The Color Trails Test measures sustained attention and sequencing. For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Cognitive Function assessed by the Wechsler Adult Intelligence Scale-III (WAIS-III) Digit Span Test | Visit 2 (Up to 2 hours)
  The Wechsler Adult Intelligence Scale-III (WAIS-III) Digit Span Test measures short-term memory, attention, and concentration. Participants will be asked to repeat 3 - 9 digits forward and 2 - 9 digits backwards.
Cognitive Function assessed by the Wechsler Adult Intelligence Scale-III (WAIS-III) Letter Number Sequence Test | Visit 2 (Up to 2 hours)
  During the Wechsler Adult Intelligence Scale-III (WAIS-III) Letter Number Sequence Test, participants will be presented with combinations of letters and numbers, (two to nine letter-number combinations). Participants will be asked to repeat each series by, first, repeating the numbers in ascending order, then the letters in alphabetical order. The test measures working memory or the ability to simultaneously recall and organize stimuli of different and similar types
Cognitive Function assessed by the Stroop Test | Visit 2 (Up to 2 hours)
  The Stroop Test measure a person's selective attention capacity and skills, as well as their processing speed ability.It is used to examine a person's executive processing abilities. The Stroop Test during brain imaging studies is used to investigate regions of the brain that are involved in planning, decision-making, and managing real-world interference
Cognitive Function assessed by the California Computerized Assessment Package (CALCAP) | Visit 2 (Up to 2 hours)
  The California Computerized Assessment Package assesses reaction times, speed of information processing, rapid visual scanning, form discrimination, brief memory and divided attention.
Self-Management assessed by the Self-care Index Heart Failure (SCHFI) | Visit 2 (Up to 2 hours)
  The Self-care Index Heart Failure (SCHFI) is a measure designed to assess self-care maintenance, management, and confidence. Participants will be asked to recall feelings of the aforementioned in the last three months.
Peak oxygen consumption assessed by the Modified Balke Test | Visit 2 (Up to 2 hours)
  Peaked oxygen consumption will be assessed by the Modified Balke Test. Participants will be asked to walk on a slightly inclined treadmill. The amount of oxygen consumed will be measured while walking for up to ten minutes.
Quality of Life assessed by the Kansas City Cardiomyopathy Questionnaire | Visit 2 (Up to 2 hours)
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gary, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia